CLINICAL TRIAL: NCT01503788
Title: Periprocedural Sedation for the Prevention of Post Dural Puncture Headache
Brief Title: Bedside Sedation for the Prevention of Post Dural Puncture Headache
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASMS-12-HS-0101-11-TLV-CTIL
Record Dates: First submitted 2012-01-01; First posted 2012-01-04 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2012-01

CONDITIONS: Post Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- periprocedural sedation with midazolam (Active Comparator): periprocedural sedation with IV midazolam 5-10 minutes before diagnostic lumbar puncture
  Interventions: Drug: Midazolam
- No intervention (No Intervention): Participants will undergo the diagnostic lumbar puncture as routinely practiced

INTERVENTIONS:
Drug: Midazolam — participants will be given Midazolam IV 10-5 minutes prior to diagnostic lumbar puncture
  Arms: periprocedural sedation with midazolam

SUMMARY:
Dural or lumbar puncture (LP), the passing of a needle into the space of the spinal cord, is a common procedure in everyday clinical practice. The most common use for LP is to measure the spinal fluid pressure and sample spinal fluid for laboratory analysis. However, it is also used for therapeutic purposes, such as administering chemotherapy or spinal anesthesia.

A notorious side effect of dural puncture is headache that ranges from mild to debilitating and may last for several days following the procedure. Among diagnosed patients, 39% experience at least 1 week of impaired ability to perform activities of daily living. The likelihood of developing a headache after dural puncture depends on a number of factors. As fluid leak is assumed to be the culprit mechanism in this headache strategies to minimize the leak seem to offer the best path to lowering the incidence of headache after diagnostic LP, the commonest clinical context of dural puncture in medical practice.

Lumbar puncture is a highly stressful event for most patients. As both pain and anxiety cause adrenergic stimulation, they also cause an increase in ICP. We believe that this mild increase in ICP, occurring before the puncture as well as during the puncture itself may exacerbate the pressure difference between the CSF space and the epidural space and so worsen the CSF leak Furthermore, this excess pressure, although mild, might cause the dural puncture hole to widen slightly and so further augment the leak and possibly even prolong it. Furthermore, the very anticipation of pain causes a rise in neurotransmitters that may cause a sensitization effect and worsen pain. This increase in adrenergic drive as well as the sensitization to pain can be effectively blunted by the periprocedural use of mild IV sedation. Benzodiazepines, with their sedative-hypnotic qualities are well suited for this task.

This study aims to test the effect of mild peri-procedural IV sedation using Midazolam on the rates of headache after diagnostic LP.

Patients undergoing a diagnostic LP will be randomized into two groups. Group 1 will undergo the procedure as routinely practiced. Group 2 will be given Midazolam IV 10-5 minutes prior to the procedure and undergo the same diagnostic procedure. All patients in the study will remain under observation in the hospital for at least 6 hours.

Patients will be evaluated for headache and specifically for headache. Clinical follow up will continue for 72 hours by administering a short questionnaire over the telephone.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* Undergoing diagnostic LP for any indication for the first time

Exclusion Criteria:

* COPD
* Any known chronic pulmonary disease
* Acute febrile illness
* Persistent headaches
* Known sensitivity to Benzodiazepines
* Current or prior substance abuse disorder
* Cognitive decline

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
rate of post dural puncture headache | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel